CLINICAL TRIAL: NCT04190563
Title: Affective and Inflammatory Reactivity to Pain in Opioid Use Disorder
Brief Title: Pain, Inflammation and Opioid Craving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, McHugh, R. Kathryn, Assistant Professor, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019P002720; R01DA045632 (NIH)
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator and data analyst will be blind to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain De-Catastrophizing (Experimental): Brief behavioral education on how to modify the interpretation of pain.
  Interventions: Behavioral: Pain De-Catastrophizing
- Pain Education (Placebo Comparator): Brief behavioral education on pain.
  Interventions: Behavioral: Pain Education

INTERVENTIONS:
Behavioral: Pain De-Catastrophizing — Experimenter-administered education and skill practice.
  Arms: Pain De-Catastrophizing
Behavioral: Pain Education — Experimenter-administered education.
  Arms: Pain Education

SUMMARY:
The goal of this study is to investigate the association between response to pain and opioid craving in people with opioid use disorder. In this study, adults with opioid use disorder will be randomized to one of two brief education sessions followed by an assessment of response to pain. Investigators will test the association between response to pain and opioid craving.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older;
* diagnosis of opioid use disorder
* chronic pain
* ability to read and provide informed consent

Exclusion Criteria:

* major psychiatric or medical condition that would interfere with participation
* current opioid withdrawal
* currently receiving opioid analgesic medication for pain
* recent history of myocardial infarction or other serious cardiovascular condition
* current peripheral neuropathy, active vasculitis or severe peripheral vascular disease
* systematic inflammatory or autoimmune disorder
* admitted to current treatment episode on an involuntary status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Craving | 30 minutes
  Investigators will assess opioid craving using the Opioid Craving Scale, a participant-reported measure of opioid craving. Investigators will measure changes in Opioid Craving Scale total scores from baseline (prior to the one-time intervention) to immediately after the intervention. This is a continuous measure that will be measured twice within this single-session experimental session. The total scale score is calculated as an average of the 3 items, with a range from 0-10, with higher scores reflecting more craving.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca K McHugh, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided